CLINICAL TRIAL: NCT03443752
Title: Comparing the Effectiveness of Shotokan-Karate vs. Tai Chi on Balance and Quality of Life in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Life Financial Movement Disorders Research and Rehabilitation Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDRC1
Record Dates: First submitted 2018-01-18; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Tai Ji

STUDY DESIGN:
Intervention Model Description: Participants will complete the experimental procedures of the present study during a 12-week training period. All participants will be asked to participate in a Shotokan-karate or Tai Chi training group. The Shotokan-karate training will involve one hour training sessions broken down into 3 components; warm-up exercises, Katas, and cool-down exercises. The protocol for Tai Chi will involve a one-hour training session which will be conducted by an instructor at the Sun Life Financial Movement Disorders and Rehabilitation Centre. All exercises will be administered by trained instructors throughout the 12-week training period. The 30-minute UPDRS assessment will be administered by Dr. Quincy Almeida,a movement disorder specialist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shotokan-Karate (Experimental): The protocol for Shotokan-karate training will involve a one hour training session which will be broken down into 3 major components. The training program will consist of warm-up exercises, katas (choreographed karate movements), and cool-down exercise.
  Interventions: Other: Shotokan-Karate
- Tai-Chi (Experimental): The protocol for Tai Chi will involve a one-hour training session which will be conducted by an instructor at the Sun Life Financial Movement Disorders and Rehabilitation Centre.The following program will be held three times per week.
  Interventions: Other: Tai-Chi

INTERVENTIONS:
Other: Shotokan-Karate — The Shotokan-Karate training program will be ran over a period of 12 weeks. Classes will be conducted 3 times per week at the Movement Disorders Rehabilitation Centre in Waterloo, Ontario. The program will be conducted by a trained professional (principal investigator), and there will be volunteers who ensure the safety and well-being of participants.
  Arms: Shotokan-Karate
Other: Tai-Chi — The Tai-Chi training program will be ran over a period of 12 weeks. Classes will be conducted 3 times per week at the Movement Disorders Rehabilitation Centre in Waterloo, Ontario. The program will be conducted by a trained professional (principal investigator), and there will be volunteers who ensure the safety and well-being of participants.
  Arms: Tai-Chi

SUMMARY:
The following study will be a comparison of balance and quality of life in Tai Chi training programs and Shotokan-Karate training programs in individuals with Parkinson's Disease. The following study will be a 12-week program which will assess whether or not Shotokan-Karate betters balance and quality of life even more than Tai Chi. Both Tai Chi and Karate will be taught by a professional instruction at the Sun Life Financial Movement Disorders and Rehabilitation Centre located in Waterloo, Ontario.

DETAILED DESCRIPTION:
Parkinson's disease is a progressive disorder of the central nervous system which affects movement. Some signs and symptoms of PD include; tremors, rigidity, gait impairments, and balance disruption. Individuals with PD experience substantially impaired balance ultimately affecting their functional abilities. With this, individuals with PD may also experience lower quality of life due to these diminished determinants. Currently, there are medications which have proven to mask the symptoms of Parkinson's such as levodopa. There are also exercise programs which have proven to improve the symptoms of Parkinson's disease such as resistance based exercises and Tai Chi.based on the proven benefits of balance and overall quality of life through Shotokan-karate training, the purpose of this study will be to compare Shotokan-karate training versus Tai Chi on balance and quality of life in individuals with Parkinson's disease. Based on the literature available on the benefits of shotokan-karate on balance and quality of life in the elderly, it is hypothesized that shotokan-karate will improve balance and quality of life due to its high intensity, increased engagement and similarities to everyday movements. If the following hypothesis is supported, the present study will allow for individuals with Parkinson's disease to engage in an exercise program that shows vast improvements in their postural stability and overall quality of life. In addition, participants will be able to engage in an exercise program which will provide them with long term benefits and they will be able to implement this in their everyday lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria involved a clinical diagnosis of Parkinson's disease, stable medication use, ability to comprehend English, ability to stand without aid and walk with or without assisted aids.

Exclusion Criteria:

* Exclusion criteria for participating in this study included any participation in current studies, which involve behavioural, cognitive or pharmacological interventions. In addition, individuals with impaired vision, impaired behavioural and cognitive abilities, and those who are unable to participate in this study due to unavailability and those with scheduling conflicts will also be apart of the exclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2018-04-03 (Estimated); Study Completion 2018-04-25 (Estimated)

PRIMARY OUTCOMES:
Change in the the Unified Parkinson's Disease Rating Scale (UPDRS) | Pre-Test (week prior), Post-Test (after 12-week training program), concluding it with a one month washout period after the completion of the study.
  Participants will be asked to complete the motor section of the Unified Parkinson's Disease Rating Scale (UPDRS-II) which will be assessed by the supervisor (Quincy J. Almeida). UPDRS-II will be assessed during the pre-testing period and the post-testing period which will be after the 12 week training program. UPDRS-II will be reassessed once again after a one month wash out period after the completion of the study. It will assess the progression of Parkinson's over the course of the exercise program and will look into how the disease has changed over time.
Change in the Parkinson's Disease Questionnaire-39 (PDQ-39). | Pre-Test (week prior), Post-Test (after 12-week training program), concluding it with a one month washout period after the completion of the study.
  PDQ-39 (Parkinson's Disease Questionnaire) is a self-reported questionnaire, which assesses a given individuals quality of life while living with Parkinson's Disease. The assessment is usually done within the ending of the designated training program. PDQ-39 assesses the experiences the participant has experienced in the training program (positive or negative), and its impact on the eight quality of life dimensions on specific areas of wellbeing in Parkinson's.
Change in the Timed Up-and-Go (TUG) Test | Pre-Test (week prior), Post-Test (after 12-week training program), concluding it with a one month washout period after the completion of the study.
  The first condiition in which balance will be measured on individuals with Parkinson's disease will be through the use of the "Timed-up-and-Go" (TUG) Test. The (TUG) Test is performed on a 4.27m long and 1.22m wide ProtoKinetics Movement Analysis Software^TM electronic walkway carpet (Zeno Walkway- Protokinetics, Haverton, PA, USA) that will capture spatiotemporal aspects of the participant's gait. The participants will begin the task by sitting on a chair placed on the Zeno Walkway. Participants will then be asked to stand up and walk to a pylon 3 meters away, then turn around at the pylon and walk back to the chair to sit down. A stopwatch will be used to record time in which it takes the participants to perform the task. The Timed Up-and-Go (TUG) Test will measure balance, ability to walk, and the risk of falls in older adults.
Change in the Gait Analysis | Pre-Test (week prior), Post-Test (after 12-week training program), concluding it with a one month washout period after the completion of the study.
  Change in Gait Analysis will be assessed through the Gait Mat which will measure an individual's step length, stride length, step variability, and the centre of pressure. Obtained results will be analyzed and calculated through a software which provides results after the completion of each trial.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886